CLINICAL TRIAL: NCT01864499
Title: Perioperative Evaluation of Intracranial Hypertension by Ultrasound Measurement of Variations in the Diameter of the Sheath of the Optic Nerve in the Excision of a Tumor or Biopsy Supratentorial Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DINO-NEURO
Record Dates: First submitted 2013-05-14; First posted 2013-05-29 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Supratentorial Brain Tumor

ARMS (2):
- Tumor Resection (Experimental)
  Interventions: Procedure: ultrasound measurement of variations in the diameter of the sheath of the optic nerve
- Biopsy Brain Tumor (Active Comparator)
  Interventions: Procedure: ultrasound measurement of variations in the diameter of the sheath of the optic nerve

INTERVENTIONS:
Procedure: ultrasound measurement of variations in the diameter of the sheath of the optic nerve — pre-and postoperative optic nerve and J2 and J5 for all patients

SUMMARY:
Neurosurgery for supratentorial brain tumor is frequently associated with preoperative intracranial hypertension. The evaluation of intracranial pressure is available noninvasively by measuring the diameter of the optic nerve sheath ultrasound.

The evaluation of intracranial pressure by measuring the DNO in perioperative is not described in the literature. The investigators propose a pilot study to assess intracranial pressure perioperative surgery for supratentorial brain tumor. The investigators consider a diameter of the optic nerve sheath as normal and predictive of intracranial pressure below 20 mm Hg when less than 5.7 mm (on the average of two measurements on each eye). DNO the normal healthy adult unanesthetized is 5 mm.

The main objective of the study is to compare the mean change in diameter of the optic nerve between the postoperative and D2 between groups of patients undergoing resection of a brain tumor and patients undergoing biopsy brain tumor.

Pilot Study: Prospective, single-center, controlled, non-randomized, the number of patients is estimated according to the recruiting capabilities of neurosurgery for this type of patient in the institution, A total of 40 patients: 20 patients Tumor Resection, control group: 20 patients Biopsy Brain Tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized for surgery of intracerebral tumors in the study group.
* Hospitalized for a biopsy of intracerebral tumor lesion in the control group.

Exclusion Criteria:

* Age <18 years
* Enucleation Prohibited to the achievement of an ocular ultrasound
* Hypersensitivity to gel
* Eye Wound
* Massive facial fracture
* Skin Infection Site

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Difference in mean changes that the sheath of postoperative optic nerve | 2 days
  Difference in mean changes that the sheath of postoperative optic nerve and J2 between groups of patients undergoing resection of brain tumor patients undergoing biopsy for brain tumor

SECONDARY OUTCOMES:
Difference in diameter of the sheath of the pre-and postoperative optic nerve | 5 days
  Difference in diameter of the sheath of the pre-and postoperative optic nerve and J2 and J5 for all patients undergoing resection of brain tumor patients undergoing biopsy for brain tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand DEBAENE, Principal Investigator — Poitiers University Hospital